CLINICAL TRIAL: NCT06717711
Title: Low-Intensity Extracorporeal Shockwave Therapy on Penile Rehabilitation After Robot-assisted Surgical Treatment of Genitourinary Cancers
Acronym: RCT_LiESWT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Principal Investigator, Giuseppe SImone, MD, Regina Elena Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PNRR-MCNT2-2023-12377570
Record Dates: First submitted 2024-11-30; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Prostate Carcinoma; Erectile Function; Genito Urinary Cancer
Keywords: prostate cancer; erectile function; rehabilitation; genitourinary cancers
MeSH Terms: conditions — Prostatic Neoplasms; Urogenital Neoplasms | interventions — Phosphodiesterase 5 Inhibitors; Tadalafil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PDE5i + LiESWT (Experimental): Patients receiving LiESWT plus early introduction of PDE5i
  Interventions: Device: Low-intensity Extracorporeal Shock Wave Therapy (LiESWT); Drug: PDE5 inhibitor (tadalafil)
- PDE5i alone (Active Comparator): Control group, patients receiving PDE5i alone
  Interventions: Drug: PDE5 inhibitor (tadalafil)

INTERVENTIONS:
Device: Low-intensity Extracorporeal Shock Wave Therapy (LiESWT) — LiESWT will be performed with PiezoWave2 from Richard Wolf and ELvation® Medical. In a single session 12,000 shocks with an energy flux density of 0.16 mJ/mm2 will be applied (4,000 over the crura of the penis and 8,000 to the penil shaft). The penis is placed in a dedicated penile holder, stretched, and shockwaves are administered with a linear therapy source (applicator) using the linear shockwave tissue coverage (LSTC-ED®) technique which makes it possible to administer shockwaves homogenously to all of the erectile tissue.
  Arms: PDE5i + LiESWT
Drug: PDE5 inhibitor (tadalafil) — Phosphodiesterase-5 (PDE5) inhibitors

SUMMARY:
This prospective randomized controlled trial (RCT) is designed to provide high level evidence on the efficacy of Low-intensity Extracorporeal Shock Wave Therapy (Li-ESWT) in the treatment of post-Robot-Assisted (RA) Radical Prostatectomy (RP) erectile dysfunction (ED) in addition to PDE5 inhibitors (PDE5i) versus PDE5i alone. Our hypothesis is that early andrological rehabilitation that combines Li-ESWT and PDE5i could lead to faster and better recovery of valid erections for intercourse, with a greater rate of postoperative International Index of Erectile Function-5 (IIEF-5) compared to patients receiving PDE5i alone.

DETAILED DESCRIPTION:
Background / State of Art ED is a common complication after radical prostatectomy, with a prevalence ranging from 40% to 80% of patients 1,2.

This considerable variability depends on the degree (intrafascial vs interfascial) and laterality (unilateral vs bilateral) of nerve sparing performed, as well as the surgical approach.

There is still paucity of high-level evidences in terms of impact of surgical approach on postoperative outcomes after RP. Considering the same surgical approach, technique, surgeon experience, patient age and preoperative erectile function remain the main predictors of postoperative sexual function.

In this context rehabilitation is still debatable and there is a lack of clear recommendations regarding the use of PDE5i and other forms of therapy. However, a multi-centre double blind RCT (n = 423) in men aged < 68 years, with normal pre-treatment erectile function undergoing either open, conventional or robot-assisted laparoscopic nerve-sparing RP, tadalafil (5 mg) once per day improved participants EPIC (Expanded Prostate Cancer Index Composite) sexual domain-scores (least squares mean difference +9.6, 95% CI: 3.1-16.0) when compared to 20 mg 'on demand' or placebo at 9 months of follow-up 3. As a result, there has been a trend toward early use of PDE5i after RP as demonstrated in some studies 4.

Hypothesis and specific aims Hypothesis and Significance The use of nerve-sparing techniques during robotic surgery has been shown to improve recovery of erectile function. However, some patients still experience ED after undergoing bilateral nerve-sparing RARP. Possible causes can be the mechanical stretching or thermal damage to cavernous nerves, ischemic injuries or local inflammation caused by surgery itself 5. Moreover, after surgery this condition could be exacerbated by an increased fibrosis and decreased elasticity of the erectile tissue in the corpora cavernosa.

Current sexual rehabilitation is essentially based on PDE5i which have been shown to increase levels of cyclic GMP in penile smooth muscle cells, preserving smooth muscle content and reducing corpora cavernosa fibrosis 6,7. At the same time, the use of vacuum erection devices, intraurethral suppositories and intracavernous injections do not guarantee an optimal penile rehabilitation after RP 8.

In this scenario, LiESWT has been recently introduced, showing promising results 9,10. It differs from other ED treatments, due to its action on the underlying pathophysiology of ED 11, offering a local remodelling of the erectile tissue 12.

Different types of energies can be used for LiESWT. The electro-hydraulic or electromagnetic generator deliver sound waves directed to the corpora cavernosa and crura, at an energy density of around 0.09 mJ/mm². Another source of energy used for LiESWT is the piezo shockwave therapy. Piezo-ceramic elements are geometrically arranged on a concave surface so that when they are excited simultaneously by a brief, high-voltage pulse, they expand by a few micrometers to generate a pressure pulse. The piezo elements are precisely aligned so that each pressure pulse generated focuses in a specific area. This precise focusing of the pulse creates a shockwave at the point of focus. The piezo shockwave's "direct focusing" technology eliminates the need for additional reflectors, resulting in a compact therapy source design and a precise and well-defined focal zone. The virtually painless therapy is quiet and energy levels can be freely adjusted with almost no adverse effect on the size of the focal zone. Extracorporeal shockwaves are mechanical stressors capable of inducing biochemical changes in living tissue; at a molecular level these changes can influence gene expression in cells and, if used selectively, can produce specific reactions in tissue. This process is referred to as mechanotransduction. The therapy was first tested for vasculogenic ED in 2010 by Vardi et al. due to its potential to promote neovascularization in the myocardium 13,14. LiESWT has also been recognized to increase nitric oxide synthesis in penile tissue and supports stem cell proliferation 15. Multiple meta-analyses suggested that LiESWT is an effective treatment for ED, resulting in an improvement in the erectile function domain scores of IIEF-5, playing a significant role not only in vasculogenic ED (neoangiogenesis) but also in neurogenesis 16,17.

However, despite the promising results, there is still a lack of high-level evidences on the use of LiESWT for ED, especially in the specific setting of postoperative rehabilitation after RP.

Our hypothesis is that LiESWT in addition to PDE5i administration could improve sexual rehabilitation with faster recovery of valid erection and higher IIEF-5 scores in the short and medium-term follow-up.

OBJECTIVES:

Primary Objective

• To investigate the impact of LiESWT in combination with early PDE5i administration versus early PDE5i alone on the penile rehabilitation of erectile dysfunction (ED) after RARP.

ED remains a significant issue after radical prostatectomy, with some of the most reliable data on patient-reported outcome measures (PROMs), including erectile function, coming from the Prostate Testing for Cancer and Treatment (ProtecT) trial. The worst trend over time was observed in the RP group, with only 21% of patients reporting erections firm enough for intercourse after 3 years, and 17% after 6 years 18. However, data regarding optimal postoperative rehabilitation of ED are still limited. The International Index of Erectile Function short form (IIEF-5) questionnaire is the recognized tool for evaluating erectile function both preoperatively and during follow-up.

The primary endpoint of this study is to determine if the difference in the final mean IIEF-5 score at last follow-up, favours the use of LiESWT in combination with PDE5i compared to early PDE5i alone for penile rehabilitation after RARP, with a minimum clinically important difference (MCID) of at least 4 points 19.

Secondary Objectives

* To compare the rate of patients who achieve orgasm and their erectile hardness score (EHS) at the final follow-up.
* To evaluate the impact of LiESWT on continence status.
* To report any adverse effects and classify them according to the Clavien Dindo classification 20.
* To compare health-related quality of life (HRQoL) outcomes at 3-, 6- and 12-months (mo) follow-up post-surgery.

Subgroup analysis An exploratory subgroup analysis will be conducted to evaluate the efficacy of LiESWT for the treatment of ED also in patients at intermediate risk PCa and in patients undergoing radical cystectomy.

STUDY DESIGN Prospective randomized controlled trial (RCT) designed to provide high level evidences describing the role of LiESWT plus early introduction of PDE5i vs early PDE5i alone on penile rehabilitation of ED after RARP.

STUDY POPULATION

Inclusion criteria:

* Patients aged ≤75 yrs;
* PSA <10 ng/mL
* Prostate Cancer ISUP grade ≤2 and cT≤2 at prostate biopsy
* undergoing nerve sparing RARP;
* preoperative IIEF-5 score ≥ 17;
* First PSA (45d after surgery) <0.1
* Prostate Cancer ISUP grade ≤2 pT<3b and at final pathology
* ≥ 18 yrs old;
* compliants patients able to follow the study protocol and fill in IIEF-5 scores and EORTC quality of life questionnaires;
* patients able to provide a written informed consent for the trial.

Exclusion criteria:

* anaesthesiologic contraindications to robotic surgery
* patients submitted to pelvic radiotherapy or androgen deprivation
* patients reporting major postoperative complications (CD≥3)
* cardiovascular contraindications to PDE5i medical treatment

Methodologies All patients for whom eligibility criteria have been verified will be enrolled and randomized by the Promoter.

Then, patients will be randomized into:

* GROUP 1 (LiESWT + PDE5i): LiESWT plus early introduction of PDE5i
* GROUP 2 (PDE5i alone): control group, PDE5i alone with on a covariate adaptive randomization process based on the following variables: Age (≥ 65 vs < 65), BMI (≥ 30 vs <30), ASA score (1-2 vs 3-4) and preoperative IIEF-5 (17-21 vs 22-25).

Patients were allocated 1:1 in each group. RARP will be performed according to EAU guidelines 21.

ASSESSMENTS Both arms will start tadalafil at a dose of 5mg/day right after the removal of the transurethral catheter, which occurs between the 7th and 10th postoperative days. All patients will receive 5 mg tadalafil tablets (7 per week), which will be dispensed weekly at each follow-up visit. Patients will be monitored for continence status (measured by pads/days), sexual function (IIEF-5 and EHS scores), and possible adverse events.

Forty-five days (45d) after surgery, the first measure of PSA will be performed.

If PSA results <0.2 ng/ml patients will be randomized. The LiESWT (6-week period) will begin one week after PSA evaluation (52d after surgery). LiESWT will be performed with PiezoWave2 from Richard Wolf and ELvation® Medical. In a single session 12,000 shocks with an energy flux density of 0.16 mJ/mm2 will be applied (4,000 over the crura of the penis and 8,000 to the penil shaft). The penis is placed in a dedicated penile holder, stretched, and shockwaves are administered with a linear therapy source (applicator) using the linear shockwave tissue coverage (LSTC-ED®) technique which makes it possible to administer shockwaves homogenously to all of the erectile tissue. Specific adverse effects that could be related to LiESWT, such as hematomas, local pain, and neuropraxia, will be assessed, classified, and recorded. Therefore, at the last follow-up, 94 days after surgery (3mo after surgery) the final IIEF-5 and EHS scores will be assessed. Afterwards, IIEF-5 and EHS scores will be collected 6 and 12 mo after surgery.

After 1 yr from surgery both groups will be asked to stop PDE5i for 2 weeks (washout period) and then IIEF-5 and EHS score will be collected without PDE5i treatment.

Each treatment will be performed in accordance with the most recent scientific evidence and European guidelines, according to oncologic departments; adverse events will be managed according to normal clinical practice.

Erectile function and HRQoL assessment Erectile function will be assessed using IIEF-5 and EHS scores, pre- and postoperatively. HRQoL will be tested before surgery and at 3-, 6- and 12-months (mo) follow-up evaluation through a self-administered validated questionnaire (EORTC-QLQ-C30 and QLQ-BLM30).

CLINICAL DATA

The following data will be collected and analysed for each patient:

* demographic data (gender, age, etc.)
* clinical and pathologic data [BMI, ASA score, haemoglobin, clinical and pathologic TNM stage, renal function (eGFR)]
* HRQoL and erectile function data

SAMPLE SIZE AND STATISTICAL CONSIDERATION According to previous studies, 4-points of difference between the final IIEF-5 means is the minimal clinically important difference (MCID) in the EF domain of the IIEF-5 scale 19. Therefore, considering a standard deviation of 9 (calculated on a previous pilot study), a power of 0.80 and α (2-sided) of 0.05, a sample size of 158 patients (79 for each cohort) is needed to test our hypothesis.

The continuous data as mean and standard deviation or median and range will be reported. Binary data will be reported as frequency and percentage values. ANOVA with repeated measures will be used for estimate primary endpoint. Student's paired t-test will be used to compare mean values, when appropriate. A p-value ≤ 0.05 will be considered statistically significant. The statistical analysis program SPSS V21 (SPSS Inc., Chicago, IL) will be used.

RANDOMIZATION Participants will be randomly assigned to group 1 or 2, based on a computer-generated randomization schedule prepared before the study by the Promoter.

Randomization is centralized and will be generated by an independent group of the promoter.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≤75 yrs;
* PSA <10 ng/mL
* Prostate Cancer ISUP grade ≤2 and cT≤2 at prostate biopsy
* undergoing nerve sparing RARP;
* preoperative IIEF-5 score ≥ 17;
* First PSA (45d after surgery) <0.1
* Prostate Cancer ISUP grade ≤2 pT<3b and at final pathology
* ≥ 18 yrs old;
* compliants patients able to follow the study protocol and fill in IIEF-5 scores and EORTC quality of life questionnaires;
* patients able to provide a written informed consent for the trial.

Exclusion Criteria:

* anaesthesiologic contraindications to robotic surgery
* patients submitted to pelvic radiotherapy or androgen deprivation
* patients reporting major postoperative complications (CD≥3)
* cardiovascular contraindications to PDE5i medical treatment

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2024-08-31 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Erectile Function | From enrollment to 1 year after treatment
  To investigate the impact of LiESWT in combination with early PDE5i administration versus early PDE5i alone on the penile rehabilitation of erectile dysfunction (ED) after RARP

SECONDARY OUTCOMES:
Urinary Continence | From enrollment to 1 year after treatment
  To evaluate the impact of LiESWT on continence status.
Adverse effects | From enrollment to 1 year after treatment
  To report any adverse effects and classify them according to the Clavien Dindo classification
Health Related Quality of Life | From enrollment to 1 year after treatment
  To compare health-related quality of life (HRQoL) outcomes at 3-, 6- and 12-months (mo) follow-up post-surgery

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - IRCCS "Regina Elena" National Cancer Institute, Rome, RM
  - IRCCS "Fondazione G. Pascale" National Cancer Institute, Naples

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mottet N, van den Bergh RCN, Briers E, Van den Broeck T, Cumberbatch MG, De Santis M, Fanti S, Fossati N, Gandaglia G, Gillessen S, Grivas N, Grummet J, Henry AM, van der Kwast TH, Lam TB, Lardas M, Liew M, Mason MD, Moris L, Oprea-Lager DE, van der Poel HG, Rouviere O, Schoots IG, Tilki D, Wiegel T, Willemse PM, Cornford P. EAU-EANM-ESTRO-ESUR-SIOG Guidelines on Prostate Cancer-2020 Update. Part 1: Screening, Diagnosis, and Local Treatment with Curative Intent. Eur Urol. 2021 Feb;79(2):243-262. doi: 10.1016/j.eururo.2020.09.042. Epub 2020 Nov 7. PMID 33172724
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Donovan JL, Hamdy FC, Lane JA, Mason M, Metcalfe C, Walsh E, Blazeby JM, Peters TJ, Holding P, Bonnington S, Lennon T, Bradshaw L, Cooper D, Herbert P, Howson J, Jones A, Lyons N, Salter E, Thompson P, Tidball S, Blaikie J, Gray C, Bollina P, Catto J, Doble A, Doherty A, Gillatt D, Kockelbergh R, Kynaston H, Paul A, Powell P, Prescott S, Rosario DJ, Rowe E, Davis M, Turner EL, Martin RM, Neal DE; ProtecT Study Group*. Patient-Reported Outcomes after Monitoring, Surgery, or Radiotherapy for Prostate Cancer. N Engl J Med. 2016 Oct 13;375(15):1425-1437. doi: 10.1056/NEJMoa1606221. Epub 2016 Sep 14. PMID 27626365
- [Background] Lin G, Reed-Maldonado AB, Wang B, Lee YC, Zhou J, Lu Z, Wang G, Banie L, Lue TF. In Situ Activation of Penile Progenitor Cells With Low-Intensity Extracorporeal Shockwave Therapy. J Sex Med. 2017 Apr;14(4):493-501. doi: 10.1016/j.jsxm.2017.02.004. Epub 2017 Mar 1. PMID 28258952
- [Background] Rosen RC, Allen KR, Ni X, Araujo AB. Minimal clinically important differences in the erectile function domain of the International Index of Erectile Function scale. Eur Urol. 2011 Nov;60(5):1010-6. doi: 10.1016/j.eururo.2011.07.053. Epub 2011 Jul 30. PMID 21855209
- [Background] Tara S, Miyamoto M, Takagi G, Kirinoki-Ichikawa S, Tezuka A, Hada T, Takagi I. Low-energy extracorporeal shock wave therapy improves microcirculation blood flow of ischemic limbs in patients with peripheral arterial disease: pilot study. J Nippon Med Sch. 2014;81(1):19-27. doi: 10.1272/jnms.81.19. PMID 24614391
- [Background] Vardi Y, Appel B, Jacob G, Massarwi O, Gruenwald I. Can low-intensity extracorporeal shockwave therapy improve erectile function? A 6-month follow-up pilot study in patients with organic erectile dysfunction. Eur Urol. 2010 Aug;58(2):243-8. doi: 10.1016/j.eururo.2010.04.004. Epub 2010 May 6. PMID 20451317
- [Background] Becker M, Goetzenich A, Roehl AB, Huebel C, de la Fuente M, Dietz-Laursonn K, Radermacher K, Rossaint R, Hein M. Myocardial effects of local shock wave therapy in a Langendorff model. Ultrasonics. 2014 Jan;54(1):131-6. doi: 10.1016/j.ultras.2013.07.005. Epub 2013 Jul 12. PMID 23896623
- [Background] Rassweiler JJ, Knoll T, Kohrmann KU, McAteer JA, Lingeman JE, Cleveland RO, Bailey MR, Chaussy C. Shock wave technology and application: an update. Eur Urol. 2011 May;59(5):784-96. doi: 10.1016/j.eururo.2011.02.033. Epub 2011 Feb 23. PMID 21354696
- [Background] Chung E, Cartmill R. Evaluation of clinical efficacy, safety and patient satisfaction rate after low-intensity extracorporeal shockwave therapy for the treatment of male erectile dysfunction: an Australian first open-label single-arm prospective clinical trial. BJU Int. 2015 Apr;115 Suppl 5:46-9. doi: 10.1111/bju.13035. PMID 25828173
- [Background] Abu-Ghanem Y, Kitrey ND, Gruenwald I, Appel B, Vardi Y. Penile low-intensity shock wave therapy: a promising novel modality for erectile dysfunction. Korean J Urol. 2014 May;55(5):295-9. doi: 10.4111/kju.2014.55.5.295. Epub 2014 May 12. PMID 24868332
- [Background] Teloken P, Mesquita G, Montorsi F, Mulhall J. Post-radical prostatectomy pharmacological penile rehabilitation: practice patterns among the international society for sexual medicine practitioners. J Sex Med. 2009 Jul;6(7):2032-8. doi: 10.1111/j.1743-6109.2009.01269.x. Epub 2009 Apr 23. PMID 19453918
- [Background] Hatzichristou D, d'Anzeo G, Porst H, Buvat J, Henneges C, Rossi A, Hamidi K, Buttner H. Tadalafil 5 mg once daily for the treatment of erectile dysfunction during a 6-month observational study (EDATE): impact of patient characteristics and comorbidities. BMC Urol. 2015 Nov 12;15:111. doi: 10.1186/s12894-015-0107-5. PMID 26563171
- [Background] Corbin JD. Mechanisms of action of PDE5 inhibition in erectile dysfunction. Int J Impot Res. 2004 Jun;16 Suppl 1:S4-7. doi: 10.1038/sj.ijir.3901205. PMID 15224127
- [Background] Ficarra V, Novara G, Ahlering TE, Costello A, Eastham JA, Graefen M, Guazzoni G, Menon M, Mottrie A, Patel VR, Van der Poel H, Rosen RC, Tewari AK, Wilson TG, Zattoni F, Montorsi F. Systematic review and meta-analysis of studies reporting potency rates after robot-assisted radical prostatectomy. Eur Urol. 2012 Sep;62(3):418-30. doi: 10.1016/j.eururo.2012.05.046. Epub 2012 Jun 1. PMID 22749850
- [Background] Philippou YA, Jung JH, Steggall MJ, O'Driscoll ST, Bakker CJ, Bodie JA, Dahm P. Penile rehabilitation for postprostatectomy erectile dysfunction. Cochrane Database Syst Rev. 2018 Oct 23;10(10):CD012414. doi: 10.1002/14651858.CD012414.pub2. PMID 30352488
- [Background] Dearnaley DP, Jovic G, Syndikus I, Khoo V, Cowan RA, Graham JD, Aird EG, Bottomley D, Huddart RA, Jose CC, Matthews JH, Millar JL, Murphy C, Russell JM, Scrase CD, Parmar MK, Sydes MR. Escalated-dose versus control-dose conformal radiotherapy for prostate cancer: long-term results from the MRC RT01 randomised controlled trial. Lancet Oncol. 2014 Apr;15(4):464-73. doi: 10.1016/S1470-2045(14)70040-3. Epub 2014 Feb 26. PMID 24581940
- [Background] Sivarajan G, Prabhu V, Taksler GB, Laze J, Lepor H. Ten-year outcomes of sexual function after radical prostatectomy: results of a prospective longitudinal study. Eur Urol. 2014 Jan;65(1):58-65. doi: 10.1016/j.eururo.2013.08.019. Epub 2013 Aug 26. PMID 24007711
- [Background] Limoncin E, Gravina GL, Corona G, Maggi M, Ciocca G, Lenzi A, Jannini EA. Erectile function recovery in men treated with phosphodiesterase type 5 inhibitor administration after bilateral nerve-sparing radical prostatectomy: a systematic review of placebo-controlled randomized trials with trial sequential analysis. Andrology. 2017 Sep;5(5):863-872. doi: 10.1111/andr.12403. Epub 2017 Aug 8. PMID 28787547